CLINICAL TRIAL: NCT05154201
Title: A Multicenter, Open-label, Phase I Clinical Study: A Dose-finding and Dose Expansion Study to Evaluate ORIN1001 Monotherapy and Its Combination in Patients With Advanced Solid Malignant Tumors
Brief Title: Treatment of Patients With Advanced Solid Tumors With Oral Agent ORIN1001 and in Combination With Standard of Care.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orinove, Inc. (Industry)
Collaborators: Fosun Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ORIN1001-C1
Record Dates: First submitted 2021-10-04; First posted 2021-12-13 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-12

CONDITIONS: Effect of Drug
Keywords: anti-tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose escalation of ORIN1001 as a single agent (Experimental): Single-agent dose escalation in Chinese patients with advanced solid tumors. Nine dose groups: 100 mg, 200 mg, 300 mg, 400 mg, 500 mg, 650 mg, 900 mg, 1200 mg, and 1500 mg orally in 21-day cycles.
  A total of 27-54 evaluable patients are expected to be enrolled. However, the dose in the escalation phase is not limited to these dose groups, and the number of enrolled patients is not limited to 27-54.
  Interventions: Drug: ORIN1001
- Dose escalation of ORIN1001 in combination with Standard of Care (Experimental): ORIN1001 will be administered daily as a tablet in combination with standard of care. This arm of the study will be carried out in 8 different cancer indications, including advanced triple-negative breast cancer received ≥ 3 lines of treatment, postmenopausal ER+/HER2-advanced breast cancer received the 1 line of treatment, advanced hepatocellular carcinoma received 1/2 line of treatment, chemotherapy-naive castrate-resistant prostatic cancer, advanced pancreatic cancer received 1/2 line of treatment, platinum-resistant/refractory advanced ovarian cancer received ≥ 2 lines of treatment, non-small cell lung cancer received ≥ 2 lines of treatment, and esophageal cancer received ≥ 2 lines of treatment.
  Interventions: Drug: ORIN1001
- Dose expansion of ORIN1001 as a single agent or in combination with Standard of Care (Experimental): After the recommended phase 2 dose of single-agent ORIN1001 is determined, a single-agent efficacy expansion study for advanced esophageal cancer, as well as a single-agent efficacy expansion study for advanced solid tumors with failure of standard treatments or no effective standard treatment.
  After the recommended phase 2 dose of the combination treatment is determined, the efficacy expansion study of the combination treatment will be conducted in the corresponding 8 different indications.
  Interventions: Drug: ORIN1001

INTERVENTIONS:
Drug: ORIN1001 — Dose escalation of ORIN1001 as a single agent or in combination with standard of care. Dose expansion of ORIN1001 as a single agent or in combination with standard of care.

SUMMARY:
Dose escalation of ORIN1001 in patients with advanced solid tumors.

Dose escalation of ORIN1001 in combination with standard of care in patients with esophageal carcinoma, metastatic breast cancer, hepatocellular carcinoma, metastatic prostate cancer, pancreatic cancer, ovarian cancer and non-small cell lung cancer.

Dose expansion of ORIN1001 as a single agent or in combination with standard of care in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Dose escalation of ORIN1001 administered as a single agent in patients with advance solid tumors. ORIN1001 is administered daily as a tablet.

Dose escalation of ORIN1001 administered in combination with standard of care in patients with esophageal carcinoma, triple negative breast cancer, ER+/HER2- metastatic breast cancer, hepatocellular carcinoma, metastatic castration-sensitive prostate cancer, pancreastic cancer, ovarian cancer and non-small cell lung cancer.

Dose expansion of single agent or combination therapy with ORIN1001 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

The patients must meet all of the following conditions:

1. Male or female, ≥ 18 years of age.
2. Single-agent dose-finding period and single-agent expansion cohort of advanced solid tumors: Patients with advanced solid tumors confirmed by histology or cytology who previously failed standard treatment (including surgery, chemotherapy, radiotherapy or biological therapy) or have no effective standard treatment; dose escalation and expansion period of combination therapy: Histologically or cytologically confirmed advanced breast cancer, hepatocellular carcinoma, prostatic cancer, pancreatic cancer, ovarian cancer, non-small cell lung cancer and esophageal cancer (see the inclusion criteria of each indication for details).
3. Provide evidence of disease progression or intolerable toxicity as confirmed by the investigator or documented in the medical history before enrollment;
4. Adequate organ functions, including all the following functions: Adequate bone marrow reserve, defined as: Absolute neutrophil count (ANC) ≥ 1.0 × 109/L; lymphocytes count ≥ 0.5 × 109/L; platelet count ≥ 100 × 109/L; hemoglobin ≥ 90 g/L; liver function (except hepatocellular carcinoma cohort): Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN), ≤ 3.0 × ULN for patients with Gilbert syndrome; aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 × ULN; ALP ≤ 2.5 × ULN; AST, ALT, ALP ≤ 5 × ULN for liver cancer patients or patients concomitantly with liver metastases; INR and APTT < 1.5 × ULN (patients receiving anticoagulant therapy are required to maintain dose stability within the recent two weeks (liver cancer patients are not allowed to take anticoagulants simultaneously for patients); renal function: Creatinine < 1.5 × ULN, or normal range of serum creatinine or creatinine clearance ≥ 50ml/min/1.73m2. Creatinine clearance is calculated using the Cockroft-Gault formula. Albumin ≥ 30 g/L.
5. Known left ventricular ejection fraction (LVEF) > 50%.
6. Coagulation function: International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
7. Patients with at least one evaluable lesion (single-agent dose escalation period) and at least one measurable lesion (single-agent dose expansion and combination therapy dose-finding/expansion period) according to RECIST Version 1.1.
8. Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 1.
9. Able to understand and willing to sign an informed consent form prior to the initiation of any study procedures; patients have an expected survival of at least 3 months.
10. Females of childbearing potential must have a negative serum pregnancy test within 14 days prior to the first dose of study drug and agree to practice contraception from 30 days prior to the first dose of study drug through 30 days after the last dose of study drug; male subjects must undergo ligation surgery or agree to practice contraception from 7 days prior to the first dose through 30 days after the last dose of study drug and refuse to donate sperm; failure rate of contraception is < 1% per year, and the typical birth control measures include double-barrier contraception, condom, oral or injectable contraceptives, intrauterine device, etc.
11. Non-hematologic toxicities of prior therapy return to ≤ Grade 1 (NCI-CTCAE version 5.0), except alopecia.

Inclusion criteria specific to triple-negative breast cancer (TNBC):

1. Male or female patients with relapsed or refractory triple-negative breast cancer who have received at least 2 prior lines of therapy or who have no standard treatment or who are unable to benefit from current therapy.
2. ER-, PR-, HER2-.

ER+/HER2- breast cancer specific inclusion criteria:

1. Patients diagnosed with ER+, HER2-, postmenopausal (≥ 18 years old) advanced breast cancer who have received one line of treatment, with evidence of local recurrence or metastasis, not suitable for surgical resection or radiotherapy with the purpose of cure, without clinical indication for chemotherapy, postmenopausal women who have not received systemic treatment;

   Menopause definition:
   1. Having received bilateral oophorectomy previously;
   2. Age ≥ 60 years;
   3. Age < 60 years and amenorrhea for 12 months or more in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression, and FSH and estradiol in the postmenopausal range (serum FSH > 40 mIU/mL and estradiol < 20 pg/mL or postmenopausal range as defined by the local laboratory).
   4. If taking tamoxifen or toremifene and aged < 60 years with FSH and estradiol in the postmenopausal range (serum FSH > 40 mIU/mL and estradiol < 20 pg/mL or per the postmenopausal range defined by local laboratory).
2. Patients must have: At least one measurable lesion according to RECIST 1.1 criteria (a lesion is considered measurable if it has been treated with radiotherapy or other local-regional therapy previously and there is clear documentation of disease progression at the treatment site after therapy completion). If there is no measurable disease, there must be at least one bone lesion dominated by lytic bone lesions (patients with no measurable disease and only one lytic bone lesion who have been previously treated with radiation therapy are eligible if there is documented evidence of disease progression in the bone lesion after radiation therapy).

Hepatocellular carcinoma specific inclusion criteria:

1. Histologically or cytologically confirmed hepatocellular carcinoma.
2. Barcelona classification (BCLC) B or C, not suitable for radical therapy (transplantation, surgical resection, ablation, etc.) or local therapy (TACE).
3. Hepatic function: Child-Pugh score A.
4. Patients with HBV or HCV infection should receive antiviral therapy for 3 months before the enrollment for treatment and should continue to receive antiviral therapy during the trial.
5. Not more than 1 prior systemic therapy.

Prostatic cancer specific inclusion criteria:

1. Histologically or cytologically confirmed prostatic adenocarcinoma.
2. Candidates for abiraterone acetate therapy with documented evidence of disease progression (after castrate levels of testosterone (< 50 ng/dl or 1.7 nmol/L) is reached, with at least one of the following: ①Biochemical relapse: PSA increased three times consecutively after an interval of more than 1 week, both increases are above 50% of the low point of PSA, and PSA > 2 ng/ml. ② Radiographic progression: Appearance of new lesions, including two or more new bone metastases on bone scan, or new soft tissue lesions evaluated using RECIST criteria.
3. Surgical or medical castration to achieve testosterone levels < 50 ng/dL (1.7 nmol/L). Subjects who have not previously undergone bilateral orchiectomy must have started treatment with a luteinizing hormone-releasing hormone (LHRH) analogue at least 4 weeks prior to Cycle 1 Day 1 and must continue the treatment during the study.
4. Patients with castration-resistant prostatic cancer who have not received prior chemotherapy

Pancreatic cancer specific inclusion criteria:

1. Definite histologically or cytologically confirmed unresectable pancreatic cancer. Patients with islet cell tumors are excluded.
2. Up to 1 prior systemic therapy (5-fluorouracil (5-FU) or gemcitabine as a radiosensitizer is not counted as a line, provided that there is no sustained toxicity for at least 6 months after the last dose).
3. Patients should be asymptomatic of jaundice or have completed biliary stent implantation before the first day after the enrollment. Massive or symptomatic ascites should be evacuated before the first day. Pain symptoms should be stable and do not require adjustment of analgesic therapy before the first day of enrollment.
4. Neutrophil count≥ 1.5 × 109/L.

Ovarian cancer specific inclusion criteria

1. Histologically confirmed and documented advanced recurrent ovarian cancer, fallopian tube cancer, and primary peritoneal cancer.
2. Platinum-refractory and platinum-resistant disease must have evidence of radiographic progression of the most recent platinum-based therapy within 6 months, calculated from the date of the last platinum-based therapy dose.
3. Having received one prior line of standard treatment.

Non-small cell lung cancer specific inclusion criteria:

1. Histologically confirmed locally advanced or metastatic non-small cell lung cancer (squamous or non-squamous).
2. Patients who have previously received at least one treatment regimen for locally advanced, unresectable/inoperable or metastatic NSCLC, and can provide evidence of disease progression during or after the last treatment (platinum-based adjuvant chemotherapy and/or neoadjuvant chemotherapy or combination therapy with curative intent (such as chemoradiotherapy)) as well as relapse within 6 months can be counted as a line of therapy.
3. Metastatic/refractory disease documented by imaging (CT scan, MRI, bone scan, etc.), clinical examinations (palpable nodules), or biopsy.
4. If there is no relevant test result of EGFR-, ALK-, the test needs to be completed at a local laboratory and the result is negative.

Esophageal cancer specific inclusion criteria:

1. Pathologically confirmed locally advanced recurrent, metastatic, or unresectable advanced esophageal squamous cell carcinoma.
2. At least 1 target lesion is measured by CT scan or MRI according to RECIST 1.1 criteria.
3. Patients who have failed in at least 1 line of standard treatment.

Exclusion Criteria:

Patients who meet any of the following criteria should not be enrolled in this clinical study:

1. Patients do not meet inclusion criteria.
2. Having received monoclonal antibody, chemotherapy, radiotherapy, or other investigational therapy within 4 weeks or 5 half-lives (whichever is shorter) before the start of dosing. Having received surgery or not recovered from surgery within 2 weeks before starting dose.
3. Central nervous system metastasis or injury without a stable control (patients with stable disease for more than 3 months who have received intracranial radiotherapy，there is no need hormone therapy are allowed).
4. Spinal cord compression was not treated with surgery and/or radical radiotherapy (previously diagnosed spinal cord compression clinically symptom or stable for ≥ 3 months after treatment is allowed.
5. Leptomeningeal disease; uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage; uncontrolled tumor-related pain.
6. Patients who have not recovered from toxic reactions caused by previous anti-tumor treatment (≥ NCI-CITCAE 5.0 grade 2, except alopecia); patients with uncontrolled diabetes (patients who are receiving stable insulin regimen or hypoglycemic agent regimen and are evaluated by specialists to have a stable blood glucose control are allowed).
7. Patients with a history of coagulation disorders; patients requiring anticoagulant or antiplatelet therapy (aspirin dose ≤ 81 mg/d, orally and subcutaneous injection of low-molecular-weight heparin preventing of deep venous thrombosis is allowed).
8. The subjects have a history of malignancy other than the indication for inclusion within the past three years, with the exception of radically treated non-melanoma basal cell carcinoma of the skin or carcinoma in situ of the cervix.
9. Patients with active infection of hepatitis B or C (except patients with liver cancer) or human immunodeficiency virus (HIV) infection or active pulmonary tuberculosis or other known active and/or uncontrolled infection.
10. Patients with serious infections, including but not limited to infectious complications, bacteremia, and severe pneumonia requiring hospitalization; patients who received intravenous antibiotics within 2 weeks before enrollment (prophylactic antibiotics e.g., antibiotics for the prevention of urinary tract infection or chronic obstructive pulmonary disease are allowed).
11. Any serious uncontrollable psychological or physical illness that would impair the patient's ability to follow protocol treatment, including but not limited to:Symptomatic congestive heart failure (congestive heart failure with New York Heart Association (NYHA) class ≥ III), unstable angina pectoris, arrhythmia, autoimmune diseases, infections and mental illness.
12. Pregnant or lactating women. Any patient who gets pregnant during the trial is to be withdrawn from the study.
13. Patients who have received prior IRE1 inhibitors.

Triple negative breast cancer (TNBC) specific exclusion criteria:

1. The investigator does not recommend re-treatment with paclitaxel because of toxicity.

ER+/HER2- breast cancer specific exclusion criteria:

1. Patients have risk of life-threatening complications or organ spread in a short term.
2. Known central nervous system uncontrolled or symptomatic metastases, the leptomeningeal metastasis.
3. (Neo) adjuvant treatment with letrozole or anastrozole within 12 months

Hepatocellular carcinoma specific exclusion criteria:

1. More than 50% of liver is occupied.
2. Bile duct invasion.
3. Main portal vein branch invasion.
4. Moderate to severe ascites with symptoms.
5. HBV DNA level ≥ 500 IU/mL.
6. Patients with untreated or incompletely curable concomitant bleeding, or gastric/esophageal varices at high risk of bleeding, or bleeding events due to gastric/esophageal varices within 6 months prior to treatment of the study.
7. Hepatic encephalopathy.
8. Coadministrate anticoagulants

Prostatic cancer-specific exclusion criteria:

1. Previous exposure to cytochrome P450 (cyp) 17 (17α-hydroxylase/C17, 20-lyase) inhibitors (e.g., abiraterone acetate, Orterone).
2. Concurrent use known strong cytochrome P450 (cyp) 3a inhibitors and moderate cyp3a inhibitors. The required washout time is 2 weeks before starting study treatment.
3. Concurrent use known strong cytochrome P450 (cyp) 3a inducers or moderate cytochrome P450 (cyp) 3a inducers. Treatment washout is 5 weeks for phenobarbital and enzalutamide and 3 weeks for other agents prior to starting study treatment.
4. Any chronic medical condition requiring systemic doses of corticosteroids greater than equivalent of 10 milligrams (mg) per day of prednisone acetate

Pancreatic cancer-specific exclusion criteria:

1. The patients have a decline in ECOG, or a greater than 20% decrease in serum albumin or 10% decrease in body weight at the baseline visit or within 72 hours prior to enrollment.
2. Patients who have received gemcitabine-containing regimens as standardized adjuvant chemotherapy or chemotherapy for advanced disease previously.
3. Known hypersensitivity to gemcitabine or adjuvants.
4. The patient is receiving coumarin anticoagulants.

Ovarian cancer specific exclusion criteria:

1. Prior allergy or intolerance to liposomal doxorubicin (PLD).

Specific exclusion criteria to non-small cell lung cancer

1. Prior treat with docetaxel.
2. Patients with hypersensitivity to known docetaxel or adjuvant.
3. Pathological diagnosis of mixed small cell and non-small cell lung cancer, or carcinoid tumor.
4. Presence of peripheral neuropathy NCI-CTCAE version 5.0 > Grade 2.

Specific Exclusion Criteria to esophageal cancer:

1. Presence of peripheral neuropathy NCI-CTCAE version 5.0 > Grade 2.
2. Patients with hypersensitivity to known docetaxel or adjuvant agents (combination treatment group).
3. Patients who have received docetaxel within 1 year (combination treatment group).
4. The tumor has invaded important blood vessels or the investigator judges that the tumor is very likely to invade important blood vessels during the subsequent study and cause fatal massive hemorrhage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Assessment of tolerability | Change from baseline through completion of study
  Whole blood sample collected for Hematology evaluation
Assessment of tolerability | Change from baseline through completion of study
  whole blood sample collected for Serum clinical chemistry
Assessment of tolerability | Change from baseline through completion of study
  Urine sample collected for Urinalysis
Assessment of tolerability | Change from baseline through completion of study
  Electrocardiogram (ECG) - A 12-lead ECG will evaluate electrical cardiac intervals P, QRS, and QT.
Assessment of tolerability | Change from baseline through completion of study
  Ultrasound Cardiogram (MUGA) will evaluate a cardiac physiologic parameter.
Assessment of tolerability | Evaluated during baseline or pre-intervention and during intervention.
  ECOG performance score (Eastern Cooperative Oncology Group) will be measured by clinician. ECOG scores range from 0 to 5. 0 is fully active and 5 is death.
Assessment of tolerability | Change from baseline through completion of study
  Body weight in kilogram (kg) will be measured on a calibrated scale.
Pharmacokinetic Evaluation | Collected on Day 1 and on Day 21 or Day 28. One cycle with single agent is 21 days and one cycle in combination with chemotherapy is 28 days.
  A blood sample will be collected to determine the concentration of ORIN1001 in plasma using analysis in a clinical lab.
Assessment of tolerability | Change from baseline through completion of study
  Blood pressure, including systolic and diastolic measurements.
Assessment of tolerability | Change from baseline through completion of study
  Pulse rate
Assessment of tolerability | Change from baseline through completion of study
  Body temperature
Assessment of tolerability | Change from baseline through completion of study
  Respiration rate

SECONDARY OUTCOMES:
Assessment of Efficacy | Change from baseline through completion of study
  CT Scan to evaluation tumor growth and size over time.
Assessment of Tumor type | Predose or baseline
  Biopsy sample - tumor genotype evaluation
Biomarker evaluation | Predose or baseline and once during intervention.
  From the biopsy of the tumor sample, immunohistochemistry evaluation will be performed to evaluate expression levels of XBP1 in tumor tissue (Pharmacodynamic-PD biomarker)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Beijing Cancer Hospital and Peking University
Locations (13):
- China (13):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Jilin Cancer Hospital, Changchun
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Harbin medical University Cancer Hospital, Harbin
  - Harbin Medical University Cancer Hospital, Heilongjiang
  - The First Affiliated Hospital of Soochow University, Jiangse
  - Harbin Medical University Cancer Hospital, Jilin
  - Shandong Provincial Cancer Hospital, Jinan
  - Shandong Provincial Cancer Hospital, Shandong
  - Shanghai Pulmonary Hospital, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Zhejiang